CLINICAL TRIAL: NCT04607278
Title: Probiotics and Prebiotics as a Potential Treatment in Fibromyalgia Patients: A Randomized, Double-Blinded, Placebo-Controlled
Brief Title: The Effect of Probiotic and Prebiotic Use on Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nazlı Nur ASLAN ÇİN, PhD, Research Assistant in Department of Nutrition and Dietetics, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-08/375
Record Dates: First submitted 2020-10-17; First posted 2020-10-29 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: probiotics; prebiotics; fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: The 8-week randomized, double-blind, parallel-group, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Patients and investigators are double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Probiotic (Experimental): Oral probiotic supplementation (Pro-Probiotic) was provided by iHealth; Cromwell, USA. Each sachet included a 1×1010 CFUs dose of four viable microbial cell preparation strains: there are two strains of lactobacillus genus (Lactobacillus acidophillus L1 (2.9×109) and Lactobacillus rhamnosus liobif (2.9×109)), Bifidobacterium longum (2.9×109) and Saccharomyces boulardii (1.3×109). Each participant took a total daily dose of 4×1010 CFUs.
  Interventions: Dietary Supplement: Probiotic
- Prebiotic (Active Comparator): The prebiotic (Inulin) was made up of inulin from the chicory plant and provided by the Fibrelle (Belgium) company. Five grams packs were given to the participants in boxes. Each participant was requested to take a total daily 10 g dose.
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): It was composed of maltodextrin, and provided by the manufacturer Fibrelle; (Belgium). The prescription was similar to probiotics or prebiotics groups.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral probiotic supplementation was provided by iHealth; Cromwell, USA. Each sachet included a 1×1010 CFUs dose of four viable microbial cell preparation strains: there are two strains of lactobacillus genus (Lactobacillus acidophillus L1 (2.9×109) and Lactobacillus rhamnosus liobif (2.9×109)), Bifidobacterium longum (2.9×109) and Saccharomyces boulardii (1.3×109). Each participant took a total daily dose of 4×1010 CFUs.
  Arms: Probiotic
Dietary Supplement: Prebiotic — The prebiotic was made up of inulin from the chicory plant and provided by the Fibrelle (Belgium) company. Five grams packs were given to the participants in boxes. Each participant was requested to take a total daily 10 g dose.
  Arms: Prebiotic
Dietary Supplement: Placebo — It was composed of maltodextrin, and provided by the manufacturer Fibrelle; (Belgium). The prescription was similar to probiotics or prebiotics groups.
  Arms: Placebo

SUMMARY:
The aim of the present study is to determine the effectiveness of probiotic and prebiotic treatments in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
Fifty-three, fibromyalgia syndrome participants were randomized to receive either: 1) probiotic 4×1010 CFUs per day 2) 10 g dose prebiotic (inulin) per day or 3) placebo for 8 wk. Fibromyalgia Impact Questionnaire (FIQ), Visual Analogical Pain Scale (VAS), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Pittsburg Sleep Quality Index (PSQI) and quality of life (SF-36) were measured during the baseline, 4 weeks and 8 weeks intervention phases. Finally, the adverse effects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-65 years.
2. Signature of informed consent by the patient.
3. Patients diagnosed according to the 2010 American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia.
4. Participants should be diagnosed with fibromyalgia at least 1 year ago.

Exclusion Criteria:

1. using of antibiotic and nutritional supplements
2. being pregnant or breastfeeding
3. the presence of any allergies
4. being involved in any medical or psychological research
5. the presence of severe gastrointestinal diseases
6. psychiatric illness other than depression and anxiety.

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 8 weeks
  Fibromyalgia Impact Questionnaire (FIQ) form is a evaluate the functional status of the patients. In this scale, 10 different features are measured: physical function, well-being, not being able to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. The scale is scored range 0-100. Low scores indicated recovery except for the feeling of well-being.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 8 weeks
  VAS was used to question the severity of the whole body pain in patients. On a 10 cm long line, "0" score indicates no pain, while "10" score indicates the most severe pain.
Beck Depression Inventory (BDI) | 8 weeks
  Depressive symptoms are assessed using the Beck Depression Inventory (BDI) which includes 21 questions with four possible answers sorted according to symptom severity. A score of 0-3 is given for each question, and the total score from the scale is ranked between 0-63. If the score increases, it indicates that the severity of depressive symptoms increases.
Beck Anxiety Inventory (BAI) | 8 weeks
  Anxiety levels were measured with the 21-item Beck Anxiety Inventory (BAI). Participants were asked to report the intensity and frequency of their feeling of anxiety using a Likert-like scale from 0 (not at all) to 3 (it bothered me a lot). If the total score increases, it increases the tendency of the individual to anxiety
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  Pittsburgh Sleep Quality Index questionnaire (PSQI) is used as a subjective measure of sleep quality and disturbances of the patient's sleep. The PSQI is a 19-item self-reported questionnaire grouped into seven score components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction). The PSQI assess behavior using Likert scales from 0 to 3, and five questions rated by the bed partner, if applicable. The PSQI yields a score from 0 (good quality) to 21 (poor quality). Global Scores >5 indicate significant sleep complaints. Those with a score of ≤5 is classified as good sleepers
SF-36 Quality of Life | 8 weeks
  SF-36 can be used for many purposes, consists of 36 questions, determines the health status of the healthy individuals or patients. The 36 multi-item scale of the short form SF-36 covers 8 aspects of physical and mental health: (1) Physical functioning (PF); (2) Role physical (RF); (3). Bodily pain (BP); (4) General health (GH); (5) Vitality (VT); (6) Social functioning (SF); (7) Role emotional (RE); (8) Mental health (MH). Domains 1 to 4 of the questionnaire deal with physical aspects, while domains 5 to 8 measure psychological features. For each parameter, scores is coded, summed and transformed to a scale from 0 (the worst possible condition) to 100 (the best possible condition).

CONTACTS AND LOCATIONS:
Overall Officials: Didem Tuba Akcali, Prof Dr, Study Director — Gazi University
Locations (1):
- Ankara University, Ankara, Kecıoren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No